CLINICAL TRIAL: NCT00388154
Title: A Phase II Study of Gemcitabine and Cisplatin for Advanced or Recurrent Endometrial Cancer
Brief Title: Gemcitabine and Cisplatin for Advanced or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0823
Record Dates: First submitted 2006-10-12; First posted 2006-10-16 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Gemcitabine; Gemzar; Gemcitabine Hydrochloride; Cisplatin; Platinol-AQ; Platinol; CDDP
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Cisplatin (Experimental): Gemcitabine 900 mg/m^2 by vein (IV) over 1 hour on Day 1 and Day 8. Cisplatin 30 mg/m^2 by vein over 1 hour on Day 1 and Day 8.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — 900 mg/m^2 by vein over 1 hour on Day 1 and Day 8.
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Cisplatin — 30 mg/m^2 by vein over 1 hour on Day 1 and Day 8.
  Other Names: Platinol-AQ; Platinol; CDDP

SUMMARY:
Primary Objective:

* To estimate the antitumor activity of the combination of gemcitabine and cisplatin in patients with advanced (stage III or IV) or recurrent endometrial cancer.

Secondary Objective:

* To determine the nature and degree of toxicity of the combination of gemcitabine and cisplatin in this cohort of patients.

DETAILED DESCRIPTION:
Gemcitabine and cisplatin are drugs that are used in the treatment of many types of cancer. Each acts to kill cancer cells throughout the body.

Before treatment starts, you will have a complete physical exam, pelvic exam, blood tests (about 2-3 teaspoons), a chest x-ray, and a CT scan or MRI. Women able to have children must have a negative blood pregnancy test.

On Day 1 and Day 8, you will receive gemcitabine chemotherapy through a small tube placed in a vein over 1 hour. This will be followed by cisplatin chemotherapy given by vein over 1 hour. Before chemotherapy is given, you will receive medications to prevent nausea. You will not receive any therapy on Day 15. One course of therapy is 3 weeks long.

Routine blood tests (about 1 teaspoon) will be done weekly during treatment and before each course of therapy (every 3 weeks). A complete checkup, including a history and physical exam, pelvic exam, and routine blood tests (about 2-3 teaspoons) will also be done before each course of therapy and a month after treatment ends. CT or MRI scans will be repeated every 2 to 3 cycles and at the end of treatment. Participants who have a partial or complete response (the tumor shrinks by more than 50% or disappears completely) will have the CT or MRI repeated at least 4 weeks later to confirm the response.

You may continue to receive treatment as long as your disease remains stable or improves. Participants who experience significant side effects may be allowed to drop to a lower dose if their disease is not worse. If the disease gets worse or if intolerable side effects occur, you will be taken off study.

When you are taken off the study, a complete medical history and physical exam will be performed. Routine blood tests (about 2-3 teaspoons) will be performed. Any side effects will be monitored until they go away.

This is an investigational study. Both of the study drugs are FDA approved and commercially available, though their use together in this study is investigational. Up to 35 patients will take part in this study. Patients will be enrolled at M.D. Anderson, St. Lukes Episcopal Hospital and The Woman's Hospital of Texas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically documented primary International Federation of Gynecology and Obstetrics (FIGO) Stage III or IV or recurrent endometrial carcinoma whose potential for cure by radiation therapy or surgery alone or in combination is very poor. Pathologic documentation of the recurrence is required.
2. Patients must have measurable disease as defined in section 8, under Criteria for Response. Disease in an irradiated field as the only site of measurable disease is acceptable only if there has been clear progression since completion of radiation treatment.
3. Patients may have received an unlimited amount of prior therapy, including platinum-based therapy, but such therapies must be discontinued at least 3 weeks prior to entry on this study. At least two weeks must have elapsed from the completion of radiotherapy and the start of therapy and six weeks must have elapsed if the radiotherapy involved the whole pelvis or over 50% of the spine, provided the acute effects of radiation treatment have resolved. Hormonal therapy may be discontinued at any time prior to initiating the protocol.
4. Patients must have adequate organ function as follows: Platelets >/= 100,000/ul; Granulocytes (ANC) >/= 1,500/ul; Creatinine </= 1.5 mg/dL serum glutamate pyruvate transaminase (SGPT/ALT) </= 3 times upper limit of normal, and Bilirubin </= 1.5 times the institutional upper limit of normal.
5. Neuropathy (sensory and motor) should be less than or equal to Common Toxicity Criteria for Adverse Effects (CTCAE) grade 1.
6. Patients must have a Zubrod Performance Status of 0, 1, or 2.
7. Patients must have signed an approved informed consent.
8. Patients must have recovered from effects of recent surgery or radiotherapy. They should be free of significant infection.

Exclusion Criteria:

1. Patients previously treated with gemcitabine.
2. Patients with a concomitant malignancy, other than non-melanoma skin cancer.
3. Patients with papillary serous or clear cell carcinoma of the endometrium, or patients with malignant mixed mullerian tumor of the uterus.
4. Patients with a prior malignancy who have been disease-free for less than 5 years.
5. Patients with concomitant medical illness such as serious uncontrolled infection, uncontrolled angina or serious peripheral neuropathy which, in the opinion of the treating physician, make the treatments prescribed on the study unreasonably hazardous for the patient.
6. Patients with renal dysfunction, chronic or acute kidney disease, or renal failure which, in the opinion of the treating physician, would make the treatments prescribed on the study unreasonably hazardous for the patient.
7. Patients whose circumstances will not permit study completion or adequate follow-up.
8. Patients who have no measurable disease.
9. Patients with a life expectancy of less than 3 months.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jubilee Brown, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - St. Lukes Episcopal Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 20, 2004 to December 19, 2008. All recruitment done within medical clinic settings at MD Anderson Cancer Center, St. Luke's Episcopal Hospital and The Woman's Hospital of Texas.
Groups:
- Gemcitabine + Cisplatin: Gemcitabine 900 mg/m^2 and Cisplatin 30 mg/m^2 by vein (IV) over 1 hour on Day 1 and Day 8.
Period: Overall Study
Arm/Group | Gemcitabine + Cisplatin
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One participant of the 21 enrolled was not evaluable for response or toxicity after transitioning to comfort care without completing the first treatment cycle.
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 75]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Zubrod performance status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status (PS) performed at baseline. PS described as 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; etc.
  participants
    0 | 15
    1 | 6
Tumor Grade [Number; unit: participants] — Endometrioid cancer grade based on how much cancer forms glands that look similar to glands found in normal, healthy endometrium. In lower-grade cancers, more of the cancerous tissue forms glands while higher-grade cancers have more of the cancer cells arranged in a disorganized way and do not form glands: Grade 1 tumors: 95%/> of cancerous tissue forming glands; Grade 2: 50% - 94% cancerous tissue form glands; and Grade 3 tumors have less than half of cancerous tissue forming glands. The higher grade, the more aggressive the cancer.
  participants
    Grade 1 | 1
    Grade 2 | 12
    Grade 3 | 8
International Federation of Gynecology & Obstetrics (FIGO) Disease Stage [Number; unit: participants] — Number participants with FIGO Stage III or IV or recurrent (any stage) endometrioid endometrial carcinoma. FIGO cancer staging system: IA-Tumor confined to uterus, no or < ½ myometrial invasion; IB-Tumor confined to uterus, > ½ myometrial invasion; I-Cervical stromal invasion, but not beyond uterus; IIIA-Tumor invades serosa or adnexa; IIIB-Vaginal and/or parametrial involvement; IIIC1-Pelvic node involvement; IIIC2- Para-aortic involvement; IVA-Tumor invasion bladder and/or bowel mucosa; IVB-Distant metastases including abdominal metastases and/or inguinal lymph nodes.
  participants
    III | 0
    IV | 5
    Recurrent | 16
Prior radiotherapy [Number; unit: participants] — Number of participants with prior radiotherapy treatments. Prior radiotherapy was allowed, but 2 weeks must have elapsed from its completion, and 6 weeks must have elapsed if radiotherapy involved the whole pelvis or >50% of the spine.
  participants
    No | 7
    Yes | 14
Prior chemotherapy regimens [Number; unit: participants] — Number of participants with none (0), 1, or 2 prior chemotherapy regimens; Participants may have received an unlimited number of prior chemotherapy agents, including platinum-based therapy, but therapy must have been discontinued 3 weeks before study enrollment.
  participants
    0 | 12
    1 | 6
    2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Participant Responses
Description: Response Evaluation Criteria In Solid Tumors (RECIST): Complete Response (CR): disappearance all target & nontarget lesions, absence new lesions, documented by 2 disease assessments 4 weeks apart; Partial response (PR): 30% decrease in sum longest diameter (LD) all measurable target lesions (baseline sum LDs as reference) & absence of progression of nontarget lesions or development of new, documented by 2 disease assessments 4 weeks apart. When only target lesion solitary pelvic mass measurable by physical examination but not radiography, a 50% decrease in LD required to be PR; Progressive disease (PD): 20% increase in sum LDs of target lesions (reference smallest sum of LDs at any assessment) or appearance of new lesions within 9 weeks of study entry, and unequivocal progression of existing nontarget lesions, other than pleural effusions without cytological proof of neoplastic origin within 9 weeks of enrollment; Stable disease (SD): any condition not meeting above CR, PR, or PD.
Time Frame: Responses required confirmation by imaging after 4-week+ interval following 3 week (21 day) therapy course.
Population: Participants who received one or more course(s) of chemotherapy and survived at least 4 weeks were considered evaluable for response; One participant was not evaluable.
Measure: Number; unit: participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 20
participants
  CR | 2
  PR | 8
  PD | 4
  SD | 6

2. Primary Outcome: Overall Objective Response Rate (CR + PR)
Description: Objective response (OR) defined as percentage of participants with RECIST Complete Response (CR) and Partial Response (PR), defined as CR: Disappearance all target and non-target lesions, no evidence of new lesions documented by 2 disease assessments at least 4 weeks apart. Normalization of CA-125, if elevated at baseline, is required; PR: 30% decrease in sum of longest dimensions (LD) of all target measurable lesions reference baseline sum of LD, no unequivocal progression of non-target lesions; no new lesions documented by 2 disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical examination, which is not radiographically measurable, a 50% decrease in the LD is required. 21-day cycle assessments or until either disease progression or adverse effects prohibit further treatment.
Time Frame: Responses required confirmation by imaging after 4-week+ interval following 3 week (21 day) therapy course.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine + Cisplatin
Number analyzed (Participants) | 20
percentage of participants | 50

ADVERSE EVENTS:
Time Frame: Participants who receive one or more course(s) of chemotherapy are evaluable for adverse effects regardless of subsequent survival. Course is 21 days. Overall study period: 11/4/04 to 1/1/13.
Arm/Group | Gemcitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 18/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Cisplatin (N=20)
Hypokalemia (Metabolism and nutrition disorders) | 4
Fatigue (General disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
Renal Insufficiency (Renal and urinary disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1 — Related to thrombocytopenia.
Neutropenia (Infections and infestations) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine + Cisplatin (N=20)
Allergy (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9
Anorexia (Gastrointestinal disorders) | 8
Atrial fibrillation (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Dehydration (Gastrointestinal disorders) | 2
Dermatologic effect (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Edema (Blood and lymphatic system disorders) | 4
Elevated Serum glutamic oxaloacetic transaminase (SGOT) (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 17
Fever (Infections and infestations) | 5
Hearing effect (Ear and labyrinth disorders) | 2
Hematuria (Blood and lymphatic system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Cardiac disorders) | 1
Infection (Infections and infestations) | 5
Mood alteration (Psychiatric disorders) | 9
Nausea (Gastrointestinal disorders) | 14
Neuropathy (Musculoskeletal and connective tissue disorders) | 6
Pain (abdominal/pelvic) (Musculoskeletal and connective tissue disorders) | 5
Pain (back) (Musculoskeletal and connective tissue disorders) | 4
Pain (bladder) (Renal and urinary disorders) | 1
Pain (extremity) (Musculoskeletal and connective tissue disorders) | 2
Pain (headache) (Nervous system disorders) | 8
Pain (joint) (Musculoskeletal and connective tissue disorders) | 3
Pain (neck) (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 2
Rigors (General disorders) | 5
Thrombosis (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 5
Urinary tract infection (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Neutropenia (Infections and infestations) | 8
Anemia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes